CLINICAL TRIAL: NCT03840642
Title: Examining an Adaptive Telehealth Intervention for Young Children With Autism Spectrum Disorder
Brief Title: Examining an Adaptive Telehealth Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Chicago (Other); National Institutes of Health (NIH) (NIH); Eotvos Lorand University (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Allison Wainer, Ph.D., Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORA 16122005; KL2TR002387 (NIH)
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Me (Active Comparator): Parents randomized to the Mirror Me condition will complete the 4 Mirror Me modules over a period of 5 weeks (~1 per week plus a week to practice). They will be provided with a visual guide for how to access the website. At 5 weeks, they will complete a remote parent-child interaction. Then they will be told their condition and to continue to use the website and practice what they have learned with their children.
  Interventions: Behavioral: Mirror Me
- Mirror Me Plus Remote Coaching (Experimental): Parents randomized to the Mirror Me plus remote coaching condition will complete the 4 Mirror Me modules over a period of 5 weeks (~1 per week plus a week to practice). They will be provided with a visual guide for how to access the website. At 5 weeks, they will complete a remote parent-child interaction. Then all parents in this condition will be told about the opportunity to participate in remote video teleconferences once per week for 5 weeks. Trained therapists will provide feedback to parents as they use the RIT techniques with their child at home. All sessions will follow a similar format including a discussion of accomplishments and challenges, parent practice with feedback, problem solving, and planning for the next week. Sessions will be recorded for data collection and therapist coaching fidelity. Participants will have access to Mirror Me for the duration of the research study.
  Interventions: Behavioral: Mirror Me; Behavioral: Remote Coaching

INTERVENTIONS:
Behavioral: Mirror Me — Mirror Me is a telehealth parent training intervention that teaches parents to promote their child's social imitation during play and daily routines. It uses content from Reciprocal Imitation Training (RIT), an evidence-based NDBI that teaches social imitation within affect-laden playful interactions. Mirror Me presents intervention content in four interactive modules. Program development was guided by the technology acceptance model, media richness theory, and principles of instructional design.
Behavioral: Remote Coaching — Trained therapists will provide feedback to parents as they use the RIT techniques with their child at home. All sessions will follow a similar format including a discussion of accomplishments and challenges, parent practice with feedback, problem solving, and planning for the next week
  Arms: Mirror Me Plus Remote Coaching

SUMMARY:
The purpose of this study is to explore the acceptability and effects of internet-based approaches for helping parents learn early intervention strategies (e.g., methods or tips for improving a child's behavior and development). As part of this study, families will be randomly(selected by chance like the flip of a coin) assigned to one of two different formats of an interactive telehealth program called Mirror Me. One format families complete on their own, the other involves the option to meet with a parent coach over the internet for feedback. The goal of the study is to understand how parents/caregivers and children benefit from using online programs, and to identify barriers (blocks) and facilitators (helpers) to this kind of service delivery model.

DETAILED DESCRIPTION:
Mirror Me is a telehealth parent training intervention that teaches parents to promote their child's social imitation during play and daily routines. It uses content from Reciprocal Imitation Training (RIT), an evidence-based NDBI that teaches social imitation within affect-laden playful interactions. RIT techniques include imitating the child (contingent imitation), modeling language, behavioral prompting, and natural reinforcement during child-direct activities. There is strong empirical support for the effect of individual techniques on imitation, joint attention, and language and RIT has been cited as one of only seven early intervention packages with "strong" evidence of efficacy with children < 3 with ASD or at risk for ASD. Because RIT focuses on a skill that emerges early in development and does not require language competency, it can be used with children at very young chronological, language, and developmental levels, making it an ideal early intervention. Given that RIT is meant to be used in a child's natural environment and only involves a handful of intervention techniques, it is well suited for delivery in a parent training format, with initial data supporting the effectiveness of parent training in RIT. Mirror Me presents intervention content in four interactive modules. Program development was guided by the technology acceptance model, media richness theory, and principles of instructional design. To ensure usability and acceptability, the investigators used an iterative development process with input from pilot participants. The investigators have subsequently upgraded the website to ensure mobile compatibility, user-friendly material, and enhanced assessment and monitoring capabilities. Mirror Me can be used as a standalone website or in combination with remote parent "coaching." Initial data indicate roughly one third to one half of parents learn RIT techniques from the website alone, while the rest require coaching. These data support the investigation of a stepped-care telehealth intervention, where parents use the Mirror Me website and then receive remote parent coaching, if the anticipated response to the program is not observed.

ELIGIBILITY:
Inclusion Criteria:

* a pre-existing diagnosis of ASD
* behaviorally-based caregiver concerns about ASD
* behaviorally-based physician concerns about ASD
* a positive screen on a validated ASD screening tool.
* a score of 40% or less on the Unstructured Imitation Assessment (UIA) at screening/baseline

Ages: 16 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Unstructured Imitation Assessment (UIA) | Baseline, Week 10, and Week 15
  An assessment that is used to measure a child's ability to imitate in a spontaneous, social-interactive context. A higher summed score on this assessment indicates better imitation abilities.
Change in Early Intervention Parenting Self Efficacy Scale | Baseline, Week 5, Week 10, Week 15
  Asks about the extent to which parents feel as though they have the skills and knowledge to help their child's development. A higher summed score on this scale indicates greater parental self-efficacy
Change in Parent Fidelity | Baseline, Week 5, Week 10, Week 15
  Ten minute parent-child play interactions videos that will be saved and later coded by trained research assistants who will be blinded to study condition.

SECONDARY OUTCOMES:
Change in Vineland Scales of Adaptive Functioning (3rd edition, survey form) | Baseline, Week 10, Week 15
  A survey administered to a parent or caregiver that is organized around four Behavior Domains:Communication, Daily Living Skills, Socialization, and Motor Skills.
Change in Social Communication Checklist Revised | Baseline, Week 10, Week 15
  Questionnaire that helps determine the child's level of child social communication skills.

OTHER OUTCOMES:
Change in Parenting Stress Index-Short Form | Baseline, Week 10, Week 15
  A caregiver self-report questionnaire that assesses dysfunctional parent-child dyads in three domains of parental-distress, difficult child characteristics, and dysfunctional parent-child interaction.
Change in Family Quality of Life Scale | Baseline, Week 10, Week 15
  Questionnaire used to determine family quality of life. Higher summed scores indicate greater family quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States